CLINICAL TRIAL: NCT06888258
Title: Comparative Study Between Ultrasound Guided Mid-point Transverse Process to Pleura Block And Erector Spinae Plane Block For Perioperative Analgesia In Modified Radical Mastectomy In Breast Cancer Patients
Brief Title: Compare Analgesia Between MTP Block And ESPB in MRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AP2407-201-014
Record Dates: First submitted 2025-02-23; First posted 2025-03-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients will be randomly assigned into three equal comparable groups using computer-generated random numbers in opaque closed envelopes, each of which will include 30 patients. With allocation ratio 1:1:1
  Group M (mid-point transverse process to pleura block MTP) N=3o Patients will receive Ultrasound guided mid-point transverse process to pleura block preoperative with injection of 20 ml bupivacaine 0.25%.Then patients will be transferred to operating room.
  Group E (Erector Spinae Plane Block ESB) N=3o Patients will receive Ultrasound guided erector spinae plane block with injection of 20 ml bupivacaine 0.25%. Patients will be transferred to operating room.
  Group C (control group) N=30 Patients will not receive any block. Induction will be performed by using a regimen of IV by fentanyl 1 μg/kg, Additional bolus doses of fentanyl 0.5 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector Spinae Plane block arm (Active Comparator): Group E: The block will be performed preoperatively with full aseptic precautions. The ultrasound probe will be placed on the back in a vertical orientation on the lateral side of the posterior median line to identify the transverse process of the 5th thoracic vertebra and erector spine muscle.
  A skin wheal using 3ml of 1% lidocaine will be made 2 to 3 cm superior to the superior aspect of the transducer. The puncture will be performed using the intra-plane needling technique after local anaesthesia infiltration. A 20-gauge Tuohy needle connected to a syringe containing the anesthetic mixture or saline will be advanced. When the puncture needle touch the transverse process, with no blood, gas, or cerebrospinal fluid observed on aspiration, 20 mL of 0.25% bupivacaine will be administered between the erector spine muscle and transverse process.
  Local anesthetic diffusion between the transverse process and erector spinae muscle is an indication of a successful puncture.
  Interventions: Procedure: Ultrasound guided Erector Spinae Plane block
- Mid-point Transverse Process to Pleura block arm (Active Comparator): Group M: The block will be performed preoperatively with full aseptic precautions. The ultrasound probe will be placed on the back in a vertical orientation on the lateral side of the posterior median line to identify the transverse processes of the 4th and 5th thoracic vertebrae and pleura.
  A skin wheal using 3ml of 1% lidocaine will be made 2 to 3 cm superior to the superior aspect of the transducer. Using the in plane needling technique in the space between the transverse processes of the 4th and 5th thoracic vertebrae, the puncture needle needle tip will be placed at the mid-point between the transverse process and pleura, with no blood, gas, or cerebrospinal fluid observed on aspiration, 20 mL of 0.25% bupivacaine will be administered. The local anesthetic spread will be noted in the area midway between the transverse process and pleura is an indication of a successful puncture.
  Interventions: Procedure: Ultrasound guided Mid-point to Pleura block
- Control arm (No Intervention): Patients in this arm will not receive block but they will receive Intravenous morphine

INTERVENTIONS:
Procedure: Ultrasound guided Erector Spinae Plane block — Group E: The block will be performed preoperatively with full aseptic precautions. The ultrasound probe will be placed on the back in a vertical orientation on the lateral side of the posterior median line to identify the transverse process of the 5th thoracic vertebra and erector spine muscle.
  A skin wheal using 3ml of 1% lidocaine will be made 2 to 3 cm superior to the superior aspect of the transducer. The puncture will be performed using the intra-plane needling technique after local anaesthesia infiltration. A 20-gauge Tuohy needle connected to a syringe containing the anesthetic mixture or saline will be advanced. When the puncture needle touch the transverse process, with no blood, gas, or cerebrospinal fluid observed on aspiration, 20 mL of 0.25% bupivacaine will be administered between the erector spine muscle and transverse process.
  Local anesthetic diffusion between the transverse process and erector spinae muscle is an indication of a successful puncture.
  Arms: Erector Spinae Plane block arm
Procedure: Ultrasound guided Mid-point to Pleura block — Group M: The block will be performed preoperatively with full aseptic precautions. The ultrasound probe will be placed on the back in a vertical orientation on the lateral side of the posterior median line to identify the transverse processes of the 4th and 5th thoracic vertebrae and pleura.
  A skin wheal using 3ml of 1% lidocaine will be made 2 to 3 cm superior to the superior aspect of the transducer. Using the in plane needling technique in the space between the transverse processes of the 4th and 5th thoracic vertebrae, the puncture needle needle tip will be placed at the mid-point between the transverse process and pleura, with no blood, gas, or cerebrospinal fluid observed on aspiration, 20 mL of 0.25% bupivacaine will be administered. The local anesthetic spread will be noted in the area midway between the transverse process and pleura is an indication of a successful puncture.
  Arms: Mid-point Transverse Process to Pleura block arm

SUMMARY:
This study is conducted to compare the analgesic efficacy between ultrasound guided Erector Spinae Plane block Vs midpoint transverse process to Pleura block in modified radical mastectomy surgeries

DETAILED DESCRIPTION:
Patients participants will be randomized into 3 groups:

Group M (mid-point transverse process to pleura block MTP) N=3o Patients will receive Ultrasound guided mid-point transverse process to pleura block preoperative with injection of 20 ml bupivacaine 0.25%.

Group M: The block will be performed preoperatively with full aseptic precautions. The ultrasound probe will be placed on the back in a vertical orientation on the lateral side of the posterior median line to identify the transverse processes of the 4th and 5th thoracic vertebrae and pleura.

A skin wheal using 3ml of 1% lidocaine will be made 2 to 3 cm superior to the superior aspect of the transducer. Using the in plane needling technique in the space between the transverse processes of the 4th and 5th thoracic vertebrae, the puncture needle needle tip will be placed at the mid-point between the transverse process and pleura, with no blood, gas, or cerebrospinal fluid observed on aspiration, 20 mL of 0.25% bupivacaine will be administered. The local anesthetic spread will be noted in the area midway between the transverse process and pleura is an indication of a successful puncture.

Group E (Erector Spinae Plane Block ESB) N=3o Patients will receive Ultrasound guided erector spinae plane block with injection of 20 ml bupivacaine 0.25%.

Group E: The block will be performed preoperatively with full aseptic precautions. The ultrasound probe will be placed on the back in a vertical orientation on the lateral side of the posterior median line to identify the transverse process of the 5th thoracic vertebra and erector spine muscle.

A skin wheal using 3ml of 1% lidocaine will be made 2 to 3 cm superior to the superior aspect of the transducer. The puncture will be performed using the intra-plane needling technique after local anaesthesia infiltration. A 20-gauge Tuohy needle connected to a syringe containing the anesthetic mixture or saline will be advanced. When the puncture needle touch the transverse process, with no blood, gas, or cerebrospinal fluid observed on aspiration, 20 mL of 0.25% bupivacaine will be administered between the erector spine muscle and transverse process.

Local anesthetic diffusion between the transverse process and erector spinae muscle is an indication of a successful puncture.

Group C (control group) N=30 Patients will not receive any block. Induction will be performed by using a regimen of IV by fentanyl 1 μg/kg, Additional bolus doses of fentanyl 0.5 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.

Randomization will be done by statistician and each group of the patient will revealed only when the included patient is transferred to preanesthetic room.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II.
* Undergoing modified radical mastectomy surgery.
* Body mass index (BMI) from 18.5 to 30 kg/m2

Exclusion Criteria:

* Patient refusal.
* Known allergy to local anesthetics.
* Bleeding disorders; platelets count <50,000 , prothrombin concentration < 60% or any coagulopathy disorder.
* Use of any anti-coagulants.
* Inability to provide informed consent.
* ASA III-IV.
* Neurological disorders.
* Patient with psychiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
post-operative opioid (morphine) consumption in the 1st 24 hours | 24 hours
  Total post operative morphine dosage in mg required

SECONDARY OUTCOMES:
Time to first rescue analgesia, starting after extubation. In minutes | 24 hours
  When was the first rescue analgesia given
Total dose of fentanyl required intraoperative (including induction dose) in microgram | 24 hours
  Total fentanyl dose given intraoperative
Numerical pain rating score at 15, 30, 45 and 60 min., 3,6,12 and 24 h after surgery. Score from 0 to 10 where 10 is the worst pain | 24 hours
  Pain score post operative
Change in heart rate (rate per minute) intraoperatively at 30 minutes interval in comparison to baseline reading. | 24 hours
  Change in vital data intraoperative
Change mean arterial blood pressure (mmHg) intraoperatively at 30 minutes interval in comparison to baseline reading. | 24 hours
  Change in vital data intraoperative
Heart rate (per minute) at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively | 24 hours
  Post operative vital data
Mean arterial blood pressure (mmHg) at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively | 24 hours
  Post operative vital data

CONTACTS AND LOCATIONS:
Overall Officials: Maie Kamal El-Din Helaly, MD, Study Director — National cancer institute, Cairo University
Locations (1):
- National cancer institute, Cairo University, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT06888258/Prot_SAP_000.pdf